CLINICAL TRIAL: NCT01755078
Title: Long Term Evaluation of Sevelamer HCl vs. Calcium-based Phosphate Binder in the Treatment of Hyperphosphatemia in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chugai Pharma Taiwan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPT-REN-002
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2012-12

CONDITIONS: Hemodialysis; Hyperphosphatemia; Cardiovascular Events
Keywords: Phosphate binder
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer; Calcium Carbonate; calcium acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer HCl (Experimental): Sevelamer HCl regular treatment 1-3 tablets TID
  Interventions: Drug: Sevelamer HCl
- Calcium-based binder (Active Comparator): Calcium-based phosphate binder (either CaCO3 or Ca acetate) administered 1-3 tablets TID
  Interventions: Drug: Calcium-based phosphate binder

INTERVENTIONS:
Drug: Sevelamer HCl — Non-metal phosphate binder
  Other Names: Renagel Tablets
  Arms: Sevelamer HCl
Drug: Calcium-based phosphate binder
  Other Names: Calcium carbonate; Calcium acetate
  Arms: Calcium-based binder

SUMMARY:
The study is designed to compare sevelamer vs. calcium-based phosphate binder in hemodialysis patients to achieve full-scale of medical care, including reduction of atherosclerotic risk factors, reduction of vascular access reconstruction rate, and pharmacoeconomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged between 18-70 years old
* Subject with hyperphosphatemia (5.5 - 8.5 mg/dL) at both WK(-2) and WK0
* On stable TIW hemodialysis for 3 months or longer

Exclusion Criteria:

* Patients with hypercalcemia (corrected serum calcium > 10.5 mg/dL)
* Any of the following abnormalities: ALT or AST > 3X ULN; iPTH > 1000 or < 150 pg/mL
* History of dysphagia or swallowing disorders
* History of GI motility disorder or GI bleeding within 3 months prior to entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Composite end-point of Ca, P, Ca*P within K/DOQI recommendation | 12 months

SECONDARY OUTCOMES:
Change from baseline, Ca, P, Ca*P | 12 months
Change from baseline, lipid profile | 12 months
Change from baseline, CRP | 12 months
Change from baseline, iPTH (stragified) | 12 months
Change from baseline, homocysteine, folate and Vit B12 | 12 months
CV-related event rate (OPD admission and hospitalization) | 12 months
Comparison of medical-related expenses between group | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Ching Huang, Professor, Principal Investigator — China Medical University Hospital

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Lin HH, Liou HH, Wu MS, Huang CC. Factors associated with serum fetuin-A concentrations after long-term use of different phosphate binders in hemodialysis patients. BMC Nephrol. 2016 Mar 23;17:33. doi: 10.1186/s12882-016-0245-3. PMID 27007989